CLINICAL TRIAL: NCT05168631
Title: Multicenter Retrospective Database on Prognostic and Predictive Factors in Patients With Neuroendocrine Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: LACOG 0119
Record Dates: First submitted 2021-12-20; First posted 2021-12-23 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Neuroendocrine Tumors; Carcinoma;Endocrine
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter retrospective longitudinal analytical study of patients with neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older and with histologically confirmed neuroendocrine tumors;
* Metastatic or inoperable disease;
* Patients with clinical information about the therapies received, including exclusive palliative care.

Exclusion Criteria:

* Lack of data on survival outcomes and/or details on treatments received.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older and with histologically confirmed neuroendocrine tumors; or metastatic or inoperable disease; or patients with clinical information about the therapies received, including exclusive palliative care.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-05-16 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2022

SECONDARY OUTCOMES:
Response rate per RECIST 1.1; | 2022
Progression-free survival by RECIST 1.1 from D1 of each treatment; | 2022
Symptom control time | 2022
  Improvement of symptoms and/or stabilization of radiological disease in non-functioning ENT, at the physician's discretion
Incidence of complications of the disease and/or treatments, defined by adverse events | 2022

CONTACTS AND LOCATIONS:
Locations (7):
- Brazil (6):
  - Universidade Federal do Ceará/HOSPITAL UNIVERSITARIO WALTER CANTIDIO, Fortaleza, Ceará
  - Ensino E Terapia de Inovacao Clinica Amo - Etica, Salvador, Estado de Bahia
  - Hospital Sírio Libanês Brasília, Brasília, Federal District
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Fundacao Antonio Prudente - Ac Camargo Center, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo
- Instituto Nacional de Enfermedades Neoplàsicas, Surquillo, Peru

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yao JC, Hassan M, Phan A, Dagohoy C, Leary C, Mares JE, Abdalla EK, Fleming JB, Vauthey JN, Rashid A, Evans DB. One hundred years after "carcinoid": epidemiology of and prognostic factors for neuroendocrine tumors in 35,825 cases in the United States. J Clin Oncol. 2008 Jun 20;26(18):3063-72. doi: 10.1200/JCO.2007.15.4377. PMID 18565894
- [Background] Hallet J, Law CH, Cukier M, Saskin R, Liu N, Singh S. Exploring the rising incidence of neuroendocrine tumors: a population-based analysis of epidemiology, metastatic presentation, and outcomes. Cancer. 2015 Feb 15;121(4):589-97. doi: 10.1002/cncr.29099. Epub 2014 Oct 13. PMID 25312765
- [Background] Dasari A, Shen C, Halperin D, Zhao B, Zhou S, Xu Y, Shih T, Yao JC. Trends in the Incidence, Prevalence, and Survival Outcomes in Patients With Neuroendocrine Tumors in the United States. JAMA Oncol. 2017 Oct 1;3(10):1335-1342. doi: 10.1001/jamaoncol.2017.0589. PMID 28448665
- [Background] Raj N, Valentino E, Capanu M, Tang LH, Basturk O, Untch BR, Allen PJ, Klimstra DS, Reidy-Lagunes D. Treatment Response and Outcomes of Grade 3 Pancreatic Neuroendocrine Neoplasms Based on Morphology: Well Differentiated Versus Poorly Differentiated. Pancreas. 2017 Mar;46(3):296-301. doi: 10.1097/MPA.0000000000000735. PMID 27759713
- [Background] Basturk O, Yang Z, Tang LH, Hruban RH, Adsay V, McCall CM, Krasinskas AM, Jang KT, Frankel WL, Balci S, Sigel C, Klimstra DS. The high-grade (WHO G3) pancreatic neuroendocrine tumor category is morphologically and biologically heterogenous and includes both well differentiated and poorly differentiated neoplasms. Am J Surg Pathol. 2015 May;39(5):683-90. doi: 10.1097/PAS.0000000000000408. PMID 25723112
- [Background] de M Rego JF, de Medeiros RSS, Braghiroli MI, Galvao B, Neto JEB, Munhoz RR, Guerra J, Nonogaki S, Kimura L, Pfiffer TE, de Castro G Jr, Hoff PM, Filho DR, Costa FP, Riechelmann RP. Expression of ERCC1, Bcl-2, Lin28a, and Ki-67 as biomarkers of response to first-line platinum-based chemotherapy in patients with high-grade extrapulmonary neuroendocrine carcinomas or small cell lung cancer. Ecancermedicalscience. 2017 Sep 11;11:767. doi: 10.3332/ecancer.2017.767. eCollection 2017. PMID 28955403
- [Background] Tang LH, Untch BR, Reidy DL, O'Reilly E, Dhall D, Jih L, Basturk O, Allen PJ, Klimstra DS. Well-Differentiated Neuroendocrine Tumors with a Morphologically Apparent High-Grade Component: A Pathway Distinct from Poorly Differentiated Neuroendocrine Carcinomas. Clin Cancer Res. 2016 Feb 15;22(4):1011-7. doi: 10.1158/1078-0432.CCR-15-0548. Epub 2015 Oct 19. PMID 26482044
- [Background] Crippa S, Partelli S, Belfiori G, Palucci M, Muffatti F, Adamenko O, Cardinali L, Doglioni C, Zamboni G, Falconi M. Management of neuroendocrine carcinomas of the pancreas (WHO G3): A tailored approach between proliferation and morphology. World J Gastroenterol. 2016 Dec 7;22(45):9944-9953. doi: 10.3748/wjg.v22.i45.9944. PMID 28018101
- [Background] Girardi DM, Silva ACB, Rego JFM, Coudry RA, Riechelmann RP. Unraveling molecular pathways of poorly differentiated neuroendocrine carcinomas of the gastroenteropancreatic system: A systematic review. Cancer Treat Rev. 2017 May;56:28-35. doi: 10.1016/j.ctrv.2017.04.002. Epub 2017 Apr 17. PMID 28456055
- [Background] Tang LH, Basturk O, Sue JJ, Klimstra DS. A Practical Approach to the Classification of WHO Grade 3 (G3) Well-differentiated Neuroendocrine Tumor (WD-NET) and Poorly Differentiated Neuroendocrine Carcinoma (PD-NEC) of the Pancreas. Am J Surg Pathol. 2016 Sep;40(9):1192-202. doi: 10.1097/PAS.0000000000000662. PMID 27259015
- [Background] Oberg K. Management of functional neuroendocrine tumors of the pancreas. Gland Surg. 2018 Feb;7(1):20-27. doi: 10.21037/gs.2017.10.08. PMID 29629316
- [Background] Mota JM, Sousa LG, Riechelmann RP. Complications from carcinoid syndrome: review of the current evidence. Ecancermedicalscience. 2016 Aug 8;10:662. doi: 10.3332/ecancer.2016.662. eCollection 2016. PMID 27594907
- [Background] Riechelmann RP, Weschenfelder RF, Costa FP, Andrade AC, Osvaldt AB, Quidute AR, Dos Santos A, Hoff AA, Gumz B, Buchpiguel C, Vilhena Pereira BS, Lourenco Junior DM, da Rocha Filho DR, Fonseca EA, Riello Mello EL, Makdissi FF, Waechter FL, Carnevale FC, Coura-Filho GB, de Paulo GA, Girotto GC, Neto JE, Glasberg J, Casali-da-Rocha JC, Rego JF, de Meirelles LR, Hajjar L, Menezes M, Bronstein MD, Sapienza MT, Fragoso MC, Pereira MA, Barros M, Forones NM, do Amaral PC, de Medeiros RS, Araujo RL, Bezerra RO, Peixoto RD, Aguiar S Jr, Ribeiro U Jr, Pfiffer T, Hoff PM, Coutinho AK. Guidelines for the management of neuroendocrine tumours by the Brazilian gastrointestinal tumour group. Ecancermedicalscience. 2017 Jan 26;11:716. doi: 10.3332/ecancer.2017.716. eCollection 2017. PMID 28194228
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009